CLINICAL TRIAL: NCT05812963
Title: Randomized Controlled Trial of Intravascular Ultrasound Versus Fractional Flow Reserve for Non-infarct Related Artery Lesions in Patients With Multivessel Disease and Acute Myocardial Infarction
Brief Title: IVUS Versus FFR for Non-infarct Related Artery Lesions in Patients With Multivessel Disease and Acute MI
Acronym: FRAME-AMI2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Chonnam National University (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FRAMEAMI119023
Record Dates: First submitted 2023-02-22; First posted 2023-04-14 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: ST Elevation Myocardial Infarction; Non-ST Elevation Myocardial Infarction
Keywords: ST-segment elevation MI; Fractional flow reserve; intravascular ultrasound; Multivessel disease; Complete revascularization; Non-ST Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized controlled non-inferiority trial to compare clinical outcomes between IVUS-guided PCI versus FFR-guided PCI in patients with acute MI and multivessel disease.
Who Masked: Outcomes Assessor
Masking Description: Clinical events will be independently adjudicated by Clinical Event Adjudication Committee (CEAC) who are blinded to clinical information or group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional flow reserve-guided PCI (Active Comparator): FFR measurement for non-IRA stenosis (>50% visual estimation) will be performed by continuous infusion of adenosine (140~180 ug/kg/min) or intracoronary nicorandil (2 mg bolus) injection. The FFR ≤0.80 will be targeted for PCI. In case of non-IRA stenosis >90%, we will judge FFR value of ≤0.80.
  Interventions: Diagnostic Test: FFR-guided PCI group
- Intravascular Ultrasound-guided PCI (Experimental): In IVUS-guided PCI group, the current trial evaluates clinical outcome following IVUS-guided treatment decision for revascularization of non-IRA stenosis. According to pre-defined criteria, the decision of revascularization will be made.
  Revascularization criteria in the IVUS-guided PCI group is 1) minimal lumen area (MLA) ≤ 3mm2 or 2) 3mm2 < MLA ≤4mm2 and plaque burden >70%.
  Interventions: Diagnostic Test: IVUS-guided PCI group

INTERVENTIONS:
Diagnostic Test: IVUS-guided PCI group — In IVUS-guided PCI group, the current trial evaluates clinical outcome following IVUS-guided treatment decision for revascularization of non-IRA stenosis.
  Arms: Intravascular Ultrasound-guided PCI
Diagnostic Test: FFR-guided PCI group — In FFR-guided PCI group, FFR measurement for non-IRA stenosis (>50% visual estimation) will be performed by continuous infusion of adenosine (140~180 ug/kg/min) or intracoronary nicorandil (2 mg bolus) injection. The FFR ≤0.80 will be targeted for PCI. In case of non-IRA stenosis >90%, we will judge FFR value of ≤0.80.
  Arms: Fractional flow reserve-guided PCI

SUMMARY:
The aim of the study is to compare clinical outcomes between intravascular ultrasound (IVUS)-guided treatment decision versus fractional flow reserve (FFR)-guided treatment decision for non-infarct related artery stenosis in patients with acute myocardial infarction (AMI) and multivessel disease.

DETAILED DESCRIPTION:
The treatment of choice of acute myocardial infarction (AMI) including ST-segment elevation myocardial infarction (STEMI) and non-ST segment elevation myocardial infarction (NSTEMI) is reperfusion therapy, preferably with percutaneous coronary intervention (PCI). While need of treating the infarct related artery (IRA) is obvious, need for routine revascularization of non-infarct related artery (non-IRA) has been a topic of debate until recent years. Through a number of observational studies, randomized trials and meta-analyses, the benefits of non-IRA PCI have been continuously implied, and COMPLETE trial with 4041 patients of STEMI and multivessel coronary artery disease in 2019 demonstrated superiority of complete revascularization to culprit-only PCI in terms of cardiovascular death or MI (primary end point) and cardiovascular death, MI, or ischemia-driven revascularization (co-primary end point). As such, complete revascularization of a significant non-IRA stenosis is recommended after successful PCI for IRA in patients with AMI and multivessel disease in current clinical guidelines.

Nevertheless, it has been unclear which criteria should be used to decide non-IRA PCI. Although potential significance of non-IRA lesions can be estimated by angiography, the limitation of angiographic visual assessment or quantitative coronary angiography has been well known. Various measurements are used for incremental information in addition to angiographic assessment in guiding PCI - namely, intravascular ultrasound (IVUS) and fractional flow reserve (FFR). IVUS provides anatomical information regarding the lumen, plaque, and plaque characteristics, and can optimize stent placement minimizing stent-related problems and lead to better clinical outcomes. On the other hand, FFR provides information on amount of ischemia which the stenosis in question is causing, and also improves the quality of PCI which has been demonstrated by multiple previous trials, and current practice guidelines recommend the use of FFR to determine revascularization strategy as Class IA recommendation. Recent trials evaluated comparative prognosis between FFR-guided versus angiograph-guided PCI for non-IRA in patients with acute MI and multivessel disease. FLOWER-MI trial showed comparable clinical outcome between FFR-guided versus angiography-guided PCI for non-IRA in STEMI patients at 1-year follow-up. FRAME-AMI trial showed superiority of FFR-guided PCI over angiography-guided PCI in reducing death, MI, or repeat revascularization during median 3.5 years of follow-up in patients with STEMI or NSTEMI and multivessel disease.

Although IVUS and FFR differ in underlying basic concepts, previous studies demonstrated clinical outcomes following treatment decision by IVUS and FFR was similar between the 2 groups. However, these studies mainly evaluated low-risk stable ischemic heart disease patients with intermediate stenosis, and does not reflect population with acute myocardial infarction undergoing complete revascularization. Currently, the data directly comparing the benefit of IVUS and FFR for non-IRA PCI in AMI is lacking. Considering that coronary atherosclerotic plaque in non-IRA of STEMI patients is associated with significantly higher risk of future clinical events, IVUS would have potential strength of detecting high risk plaque in non-IRA and treatment decision based on plaque characteristics. Conversely, FFR-guided treatment decision for non-IRA would detect functionally significant non-IRA stenosis and treatment decision based on functional significance would reduce unnecessary PCI, as demonstrated by previous trials.

In this regard, randomized controlled trial comparing clinical outcome following non-IRA PCI in AMI patients with multivessel disease guided by IVUS or FFR would provide valuable evidence to enhance patient's prognosis after treatment of STEMI. Therefore, FRAME-AMI 2 trial is designed to compare clinical outcomes after non-IRA PCI using either IVUS-guided or FFR-guided strategy.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 19 years of age
* Acute ST-segment elevation myocardial infarction (STEMI)

  *STEMI: ST-segment elevation ≥0.1 mV in ≥2 contiguous leads or documented newly developed left bundle-branch block
* Acute non-ST-segment elevation myocardial infarction (NSTEMI)

  *NSTEMI: NSTEMI is defined as a combination of criteria with mandated elevation of a cardiac biomarker, preferably high-sensitive cardiac troponin with at least one value above 99th percentile of the upper reference limit and at least one of the following:
  1. Symptoms of ischemia.
  2. New or presumed new significant ST-T wave changes
  3. Development of pathological Q waves on electrocardiography.
  4. Imaging evidence of new or presumed new loss of viable myocardium or regional wall motion abnormality.
  5. Intracoronary thrombus detected on angiography.
* Successful primary percutaneous coronary intervention (PCI) in < 12 h after the onset of symptoms for STEMI patients (In case of NSTEMI, PCI should be performed within 72 hours of symptom onset)
* Multivessel disease (at least one stenosis of >50% in a non-IRA ≥2.25 mm by visual estimation)
* Subject is able to verbally confirm understandings of risks, benefits and treatment alternatives of receiving invasive physiologic evaluation and PCI and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure.

Exclusion Criteria:

* Non-IRA stenosis not amenable for PCI treatment by operators' decision
* Cardiogenic shock (Killip class IV) already at presentation or the completion of IRA PCI
* Intolerance to Aspirin, Clopidogrel, Prasugrel, Ticagrelor, Heparin, or Everolimus
* Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
* Pregnancy or breast feeding
* Non-cardiac co-morbid conditions are present with life expectancy <2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Other primary valvular disease with severe degree: severe mitral regurgitation, mitral stenosis, severe aortic regurgitation, or aortic stenosis
* Unwillingness or inability to comply with the procedures described in this protocol.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2023-09-18 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient-Oriented Composite Outcome | 2 years after last patient enrollment
  a composite of death, myocardial infarction, or repeat revascularization

SECONDARY OUTCOMES:
All-cause death | 2 years after last patient enrollment
  All-cause death
Cardiac death | 2 years after last patient enrollment
  Cardiac death
Spontaneous myocardial infarction | 2 years after last patient enrollment
  Spontaneous myocardial infarction, defined by Forth Universal definition of myocardial infarction
Procedure-related myocardial infarction | 2 years after last patient enrollment
  Procedure-related myocardial infarction, defined by ARC II definition
Any revascularization | 2 years after last patient enrollment
  Any revascularization (clinically-driven or ischemia-driven)
Infarct-related artery revascularization | 2 years after last patient enrollment
  Infarct-related artery revascularization
Non-Infarct-related artery revascularization | 2 years after last patient enrollment
  Non-Infarct-related artery revascularization
Definite or probable stent thrombosis | 2 years after last patient enrollment
  Definite or probable stent thrombosis
Stroke (ischemic or hemorrhagic) | 2 years after last patient enrollment
  Stroke (ischemic or hemorrhagic)
Total procedural time | at least 1 week after index procedure
  Total procedural time (from the end of primary PCI for IRA to the completion of non-IRA PCI including amount of staged procedure)
Total fluoroscopy time | at least 1 week after index procedure
  Total fluoroscopy time (from the end of primary PCI for IRA to the completion of non-IRA PCI including amount of staged procedure)
Total amount of contrast use | at least 1 week after index procedure
  Total amount of contrast use (from the end of primary PCI for IRA to the completion of non-IRA PCI including amount of staged procedure)
Incidence of contrast-induced nephropathy | at least 1 week after index procedure
  Incidence of contrast-induced nephropathy, defined as an increase in serum creatinine of ≥0.5mg/dL or ≥25% from baseline within 48-72 hours after contrast agent exposure.
A composite of all-cause death or myocardial infarction | 2 years after last patient enrollment
  A composite of all-cause death or myocardial infarction
A composite of cardiac death or non-procedure-related myocardial infarction | 2 years after last patient enrollment
  A composite of cardiac death or non-procedure-related myocardial infarction
Angina severity by Seattle Angina Questionnaire | At 2 years from index procedure
  Angina severity by Seattle Angina Questionnaire
Quality of life by EQ-5D-5L Questionnaire | At 2 years from index procedure
  Quality of life by EQ-5D-5L Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Principal Investigator — Samsung Medical Center; Young Joon Hong, MD, PhD, Principal Investigator — Chonnam National University
Locations (2):
- South Korea (2):
  - Chonnam National University, Gwangju
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Yes
After publication of main paper, de-identified data will be shared upon reasonable requests after discussion by Executive Committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of main paper.
Access Criteria: Executive Committee will discuss to share the de-identified data upon reasonable requests.